CLINICAL TRIAL: NCT04623450
Title: The Effect of Different Macronutrients on Appetite and Satiety in Older and Younger Adults
Brief Title: Macronutrients and Satiety in Older and Younger Adults
Acronym: MACROSAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Reading (Other)
Collaborators: Ministry of National Education, Turkey (Other Government)
Responsible Party: Principal Investigator, Miriam Clegg, Lecturer, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: UREC 19/25
Record Dates: First submitted 2020-10-28; First posted 2020-11-10 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Appetitive Behavior; Gastric Emptying
Keywords: younger adults; older adults; appetite; satiety; macronutrients
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Carbohydrate Meal (Experimental): A smoothie including maltodextrin and low-fat strawberry yoghurt - 289 kcal, 61g carbohydrate, 6.7g protein, 1.9g fat.
  Interventions: Other: Smoothie
- High Fat Meal (Experimental): A smoothie including double cream and low-fat strawberry yoghurt - 312 kcal, 13.3g carbohydrate, 7g protein, 25.5g fat.
  Interventions: Other: Smoothie
- High Protein Meal (Experimental): A smoothie including whey protein and low-fat strawberry yoghurt - 307 kcal, 13.6g carbohydrate, 57g protein, 2.7g fat.
  Interventions: Other: Smoothie

INTERVENTIONS:
Other: Smoothie — Preload smoothies that are matched for taste, smell, appearance, quantity and calorie but different caloric content.

SUMMARY:
This study aims to compare the effect of meals high in protein, fat and carbohydrate but equal in energy and volume on energy intake, perceived appetite and gastric emptying in younger (<40 years) and older (> 65 years) people living in the United Kingdom (UK).

DETAILED DESCRIPTION:
To assess if increasing protein intake in older adults will have a compensatory decrease in energy intake due to protein's satiating effects.

To compare the effect of meals high in protein, fat and carbohydrate but equal in energy and volume on energy intake and perceived appetite in younger (<40 years) and older adults (>65 years).

To compare the effect of meals high in protein, fat and carbohydrate but equal in energy and volume on gastric emptying in younger (<40 years) and older adults (>65 years).

ELIGIBILITY:
Inclusion Criteria:

* either aged >65 years or <40 years
* healthy

Exclusion Criteria:

* having a disease and/or using a medication that can impact on appetite in the past three months;
* having an allergy to any of the test foods;
* disliking or cannot eat any of the test foods;
* being pregnant or breastfeeding;
* being obese (BMI > 30 kg/m2);
* being on a weight loss diet;
* smoking more than 10 cigarettes a day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-05-05 (Actual); Primary Completion 2021-06-07 (Estimated); Study Completion 2021-09-09 (Estimated)

PRIMARY OUTCOMES:
Ad-libitum meal consumption | 3 days in total
  Consumption of the ad-libitum meal is measured (g). Participants are instructed to eat until they feel comfortable full and are given 20 min to consume the meal.

SECONDARY OUTCOMES:
Ratings of appetite | 3 days in total
  Appetite are assessed using a 100 mm Visual Analogue Scales (VAS, scale 0-100).
Gastric Emptying | 3 days in total
  Gastric emptying is measured using of 13C octanoic acid breath test
Ratings of palatability | 3 days in total
  Palatability ratings are assessed using a 100 mm Visual Analogue Scales (VAS, scale 0-100).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No personal identification data will be shared. The study is not under an obligation to share data, however, it is possible that some of the individual (unliked / non-identifiable) data will be useful in a meta-analysis and, hence sharing individual participant data (IPD) will be considered.

REFERENCES:
- [Background] Deutz NE, Bauer JM, Barazzoni R, Biolo G, Boirie Y, Bosy-Westphal A, Cederholm T, Cruz-Jentoft A, Krznaric Z, Nair KS, Singer P, Teta D, Tipton K, Calder PC. Protein intake and exercise for optimal muscle function with aging: recommendations from the ESPEN Expert Group. Clin Nutr. 2014 Dec;33(6):929-36. doi: 10.1016/j.clnu.2014.04.007. Epub 2014 Apr 24. PMID 24814383
- [Background] Clarkston WK, Pantano MM, Morley JE, Horowitz M, Littlefield JM, Burton FR. Evidence for the anorexia of aging: gastrointestinal transit and hunger in healthy elderly vs. young adults. Am J Physiol. 1997 Jan;272(1 Pt 2):R243-8. doi: 10.1152/ajpregu.1997.272.1.R243. PMID 9039015
- [Background] Blundell JE, Burley VJ, Cotton JR, Lawton CL. Dietary fat and the control of energy intake: evaluating the effects of fat on meal size and postmeal satiety. Am J Clin Nutr. 1993 May;57(5 Suppl):772S-777S; discussion 777S-778S. doi: 10.1093/ajcn/57.5.772S. PMID 8475895
- [Background] Rolls BJ, Kim-Harris S, Fischman MW, Foltin RW, Moran TH, Stoner SA. Satiety after preloads with different amounts of fat and carbohydrate: implications for obesity. Am J Clin Nutr. 1994 Oct;60(4):476-87. doi: 10.1093/ajcn/60.4.476. PMID 7661908
- [Background] Clegg ME, Williams EA. Optimizing nutrition in older people. Maturitas. 2018 Jun;112:34-38. doi: 10.1016/j.maturitas.2018.04.001. Epub 2018 Apr 4. PMID 29704915
- [Background] Giezenaar C, Trahair LG, Luscombe-Marsh ND, Hausken T, Standfield S, Jones KL, Lange K, Horowitz M, Chapman I, Soenen S. Effects of randomized whey-protein loads on energy intake, appetite, gastric emptying, and plasma gut-hormone concentrations in older men and women. Am J Clin Nutr. 2017 Sep;106(3):865-877. doi: 10.3945/ajcn.117.154377. Epub 2017 Jul 26. PMID 28747330
- [Background] Appleton KM. Limited compensation at the following meal for protein and energy intake at a lunch meal in healthy free-living older adults. Clin Nutr. 2018 Jun;37(3):970-977. doi: 10.1016/j.clnu.2017.03.032. Epub 2017 Apr 7. PMID 28431774
- [Background] Beelen J, de Roos NM, de Groot LC. Protein Enrichment of Familiar Foods as an Innovative Strategy to Increase Protein Intake in Institutionalized Elderly. J Nutr Health Aging. 2017;21(2):173-179. doi: 10.1007/s12603-016-0733-y. PMID 28112772